CLINICAL TRIAL: NCT03195283
Title: A Novel In-hospital Meal Service Improves Protein and Energy Intake
Brief Title: Novel Meal Service Improves Nutritional Intake
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1805
Record Dates: First submitted 2017-06-02; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-05

CONDITIONS: Malnutrition
Keywords: meal service; protein intake; satisfaction; hospitalized patients
MeSH Terms: conditions — Malnutrition; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traditional meal service: TMS consists of three meals served by nutritional assistants throughout the day. Preference for dinner can be indicated in the morning by the individual patient from a menu list with predefined choices for meat, potatoes/rice/pasta and vegetables with various portion sizes.
  Interventions: Other: Meal service
- FoodforCare: FfC consists of a 6-meals per day service. At bedside, patients are offered one or more small protein-rich dishes from a choice of 3. Nutritional assistants play a key role in recommending and delivering these protein-rich meals and assist patient in choosing the most optimal dish, based on the patient's nutrition order in the electronic patient record.
  Interventions: Other: Meal service

INTERVENTIONS:
Other: Meal service — The type of meal service in the hospital (usual care)

SUMMARY:
This study aims to investigate whether a novel meal service FoodforCare (FfC), comprising 6-protein-rich meals a day following proactive advice from a nutritional assistant, improves dietary intake and patient satisfaction, compared to the traditional 3-meals a day service (TMS).

DETAILED DESCRIPTION:
The investigators performed a quasi experimental study at medical (Gastroenterology) and surgical (Gynecology, Urology, Orthopedics) wards. Patients were offered TMS (July 2015 - May 2016; n=326) or FfC meal service (after stepwise introduction per ward from January 2016 - December 2016; n=311). Primary outcome was the mean percentage of protein and energy intake relative to requirements, between patients receiving TMS and those receiving FfC, on the first and fourth day of full oral intake. Patient satisfaction comprised rating of the experienced quality of the food and the meal service and by means of a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking
* Aged 18 years or older
* Exclusively oral intake
* Expected hospital stay of at least 1 day

Exclusion Criteria:

* Patients with tube- or parenteral feeding
* A language barrier
* Considered to be too weak to adequately answer our questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Departments of Gastroenterology, Urology/Gynaecology and Orthopedics.
Sampling Method: Non-Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Protein intake day 1 (gram) | 1 day
  The percentage of protein intake (gram) relative to requirements (1.2 gram/kilogram bodyweight) on the first day of full oral intake.
Protein intake day 4 (gram) | 4 days
  The percentage of protein intake (gram) relative to requirements (1.2 gram/kilogram bodyweight) on the fourth day of full oral intake.
Energy intake day 1 (kcal) | 1 day
  The percentage of energy intake (kcal) relative to requirements (Harris & Benedict formula * 1.3) on the first day of full oral intake.
Energy intake day 4 (kcal) | 4 days
  The percentage of energy intake (kcal) relative to requirements (Harris & Benedict formula * 1.3) on the fourth day of full oral intake.

SECONDARY OUTCOMES:
Patients' satisfaction (food appreciation and access to food) | 3 day
  Patients completed a questionnaire on food appreciation and experiences regarding food access on the third day of full oral intake in the hospital.
Patients' satisfaction (food quality and meal service) | 3 day
  Patients completed a questionnaire in which they rated the quality of the food and the meal service (scale 0-10) on the third day of full oral intake in the hospital.
Change in nutritional status (body weight) | 4 days
  Body weight (in kg) was measured prior to meals in the morning of the first and fourth day of oral intake.
Change in nutritional status (handgrip strength) | 4 days
  Handgrip strength (in kg) was measured prior to meals in the morning of the first and fourth day of oral intake.
Nutritional status (height) | 1 day
  Height (in cm) was measured prior to meals in the morning of the first day of oral intake.
Nutritional status (malnutrition universal screening tool) | 1 day
  Malnutrition universal screening tool (MUST)) was measured prior to meals in the morning of the first day of oral intake. Weight (kg) and height (cm) will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Wanten, MD, PhD, MSc, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stratton RJ, Hackston A, Longmore D, Dixon R, Price S, Stroud M, King C, Elia M. Malnutrition in hospital outpatients and inpatients: prevalence, concurrent validity and ease of use of the 'malnutrition universal screening tool' ('MUST') for adults. Br J Nutr. 2004 Nov;92(5):799-808. doi: 10.1079/bjn20041258. PMID 15533269
- [Background] Norman K, Pichard C, Lochs H, Pirlich M. Prognostic impact of disease-related malnutrition. Clin Nutr. 2008 Feb;27(1):5-15. doi: 10.1016/j.clnu.2007.10.007. Epub 2007 Dec 3. PMID 18061312
- [Background] Kondrup J, Allison SP, Elia M, Vellas B, Plauth M; Educational and Clinical Practice Committee, European Society of Parenteral and Enteral Nutrition (ESPEN). ESPEN guidelines for nutrition screening 2002. Clin Nutr. 2003 Aug;22(4):415-21. doi: 10.1016/s0261-5614(03)00098-0. PMID 12880610
- [Background] Lucy Kok RS. Ondervoeding onderschat. De kosten van ondervoeding en het rendement van medische voeding. Amsterdam: SEO economisch onderzoek, 2014.
- [Background] Beck AM, Balknas UN, Furst P, Hasunen K, Jones L, Keller U, Melchior JC, Mikkelsen BE, Schauder P, Sivonen L, Zinck O, Oien H, Ovesen L; Council of Europe (the Committee of Experts on Nutrition, Food Safety and Consumer Health of the Partial Agreement in the Social and Public Health Field). Food and nutritional care in hospitals: how to prevent undernutrition--report and guidelines from the Council of Europe. Clin Nutr. 2001 Oct;20(5):455-60. doi: 10.1054/clnu.2001.0494. PMID 11534942
- [Background] Health Do. Essence of Care. Patient-focused benchmarks for clinical governance. Publication. London: NHS Modernisation Agency potDoH; 2003.
- [Background] van Bokhorst-de van der Schueren MA, Roosemalen MM, Weijs PJ, Langius JA. High waste contributes to low food intake in hospitalized patients. Nutr Clin Pract. 2012 Apr;27(2):274-80. doi: 10.1177/0884533611433602. Epub 2012 Feb 29. PMID 22378801
- [Background] Hiesmayr M, Schindler K, Pernicka E, Schuh C, Schoeniger-Hekele A, Bauer P, Laviano A, Lovell AD, Mouhieddine M, Schuetz T, Schneider SM, Singer P, Pichard C, Howard P, Jonkers C, Grecu I, Ljungqvist O; NutritionDay Audit Team. Decreased food intake is a risk factor for mortality in hospitalised patients: the NutritionDay survey 2006. Clin Nutr. 2009 Oct;28(5):484-91. doi: 10.1016/j.clnu.2009.05.013. Epub 2009 Jul 1. PMID 19573957
- [Background] Naithani S, Thomas JE, Whelan K, Morgan M, Gulliford MC. Experiences of food access in hospital. A new questionnaire measure. Clin Nutr. 2009 Dec;28(6):625-30. doi: 10.1016/j.clnu.2009.04.020. Epub 2009 May 27. PMID 19477558
- [Background] Wall BT, van Loon LJ. Nutritional strategies to attenuate muscle disuse atrophy. Nutr Rev. 2013 Apr;71(4):195-208. doi: 10.1111/nure.12019. Epub 2013 Feb 28. PMID 23550781
- [Background] Inspectie voor de Gezondheidszorg (IGZ). Kwaliteitsindicatoren 2014 basisset ziekenhuizen. Utrecht, The Netherlands: Ministerie van Volksgezondheid, Welzijn en Sport, 2014
- [Background] Mueller C, Compher C, Ellen DM; American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) Board of Directors. A.S.P.E.N. clinical guidelines: Nutrition screening, assessment, and intervention in adults. JPEN J Parenter Enteral Nutr. 2011 Jan;35(1):16-24. doi: 10.1177/0148607110389335. No abstract available. PMID 21224430
- [Background] Mulasi U, Kuchnia AJ, Cole AJ, Earthman CP. Bioimpedance at the bedside: current applications, limitations, and opportunities. Nutr Clin Pract. 2015 Apr;30(2):180-93. doi: 10.1177/0884533614568155. Epub 2015 Jan 22. PMID 25613832
- [Background] Flood A, Chung A, Parker H, Kearns V, O'Sullivan TA. The use of hand grip strength as a predictor of nutrition status in hospital patients. Clin Nutr. 2014 Feb;33(1):106-14. doi: 10.1016/j.clnu.2013.03.003. Epub 2013 Mar 27. PMID 23615623
- [Background] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Background] Vera Todorovic CRaME. THE 'MUST' EXPLANATORY BOOKLET. A Guide to the 'Malnutrition Universal Screening Tool' ('MUST') for Adults. UK: 2011.
- [Derived] Dijxhoorn DN, van den Berg MGA, Kievit W, Korzilius J, Drenth JPH, Wanten GJA. A novel in-hospital meal service improves protein and energy intake. Clin Nutr. 2018 Dec;37(6 Pt A):2238-2245. doi: 10.1016/j.clnu.2017.10.025. Epub 2017 Nov 9. PMID 29173893